CLINICAL TRIAL: NCT03190135
Title: Evaluation of the Build Our Kids' Success (BOKS) Before-school Physical Activity Program
Brief Title: Evaluation of the BOKS Before-school Physical Activity Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Reeboks BOKS (Unknown)
Responsible Party: Principal Investigator, Elsie Taveras, MD, Chief, Division of General Academic Pediatrics, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017P000177
Record Dates: First submitted 2017-06-09; First posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Overweight and Obesity; Affect; Physical Activity; Fitness
Keywords: Overweight; Obesity; School; Physical Activity
MeSH Terms: conditions — Overweight; Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BOKS: 2 day per week (Experimental)
  Interventions: Behavioral: BOKS: 2 day a week before-school physical activity program
- BOKS: 3 day per week (Experimental)
  Interventions: Behavioral: BOKS: 3 day a week before-school physical activity program
- Non-BOKS (No Intervention)

INTERVENTIONS:
Behavioral: BOKS: 2 day a week before-school physical activity program — Students participate in BOKS, a before-school physical activity program for 12 weeks, 2 times per week.
  Arms: BOKS: 2 day per week
Behavioral: BOKS: 3 day a week before-school physical activity program — Students participate in BOKS, a before-school physical activity program for 12 weeks, 3 times per week.
  Arms: BOKS: 3 day per week

SUMMARY:
BOKS, Build Our Kids' Success, is a before-school physical activity program that has been implemented in over 2,000 elementary and middle schools. Students participate in the program for 12 weeks, two or three mornings per week for about 1 hour per session. This study if a non-randomized control trial seeking to 1) examine the extent to which participation in the before-school BOKS program improves, health, well-being, and performance, and 2) compare the results of a two-day-per-week versus a three-day-per-week program.

ELIGIBILITY:
Inclusion Criteria:

* Participating school
* Child age 5-14 years

Exclusion Criteria:

* No valid parental consent
* Missing group assignment

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1250 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2016-05-31 (Actual); Study Completion 2016-05-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline Body Mass Index at 12 weeks | baseline, 12 weeks
  Body Mass Index (kg/m^2): calculated from height and weight
Change from baseline Body Mass Index Z-score at 12 weeks | baseline, 12 weeks
  Age- and sex- specific Body Mass Index Z-score

SECONDARY OUTCOMES:
Change from baseline 400 meter run time at 12 weeks | baseline, 12 weeks
  Time (seconds) to complete a 400 meter run
Change from baseline physical activity at 12 weeks | baseline, 12 weeks
  Days per week of physical activity
Change from baseline peer relationships at 12 weeks | baseline, 12 weeks
  PROMIS validated scale
Change from baseline positive affect at 12 weeks | baseline, 12 weeks
  PROMIS validated scale
Change from baseline life satisfaction at 12 weeks | baseline, 12 weeks
  PROMIS validated scale
Change from baseline vitality/energy at 12 weeks | baseline, 12 weeks
  Healthy Pathways Child-Report Scales
Change from baseline student engagement at 12 weeks | baseline, 12 weeks
  Healthy Pathways Child-Report Scales

CONTACTS AND LOCATIONS:
Overall Officials: Elsie Taveras, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Plymouth Public Schools, Plymouth, Massachusetts
  - Quincy Public Schools, Quincy, Massachusetts
  - Weymouth Public Schools, Weymouth, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pojednic R, Peabody S, Carson S, Kennedy M, Bevans K, Phillips EM. The effect of before school physical activity on child development: A study protocol to evaluate the Build Our Kids Success (BOKS) Program. Contemp Clin Trials. 2016 Jul;49:103-8. doi: 10.1016/j.cct.2016.06.009. Epub 2016 Jun 23. PMID 27339866
- [Derived] Whooten RC, Perkins ME, Gerber MW, Taveras EM. Effects of Before-School Physical Activity on Obesity Prevention and Wellness. Am J Prev Med. 2018 Apr;54(4):510-518. doi: 10.1016/j.amepre.2018.01.017. Epub 2018 Feb 12. PMID 29449135